CLINICAL TRIAL: NCT04885933
Title: The Impact of Sarcopenia on COPD Exacerbation Admission Outcome and Further Exacerbation Risk
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FEMH-106099-E
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Sarcopenia; COPD Exacerbation
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD exacerbation
  Interventions: Diagnostic Test: sarcopenia measurement

INTERVENTIONS:
Diagnostic Test: sarcopenia measurement — BIA for fat free muscle mass hand grasp strength

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is more prevalent and has more impact on health status because of progressive air pollution, tobacco smoking and aging society. The COPD prevalence investigation in 2013 by phone call showed at least 6% of the population with more than 40 years-old in Taiwan. It also was the 7th ranking of death causes in Taiwan then. Apart from chronic inflammation in lung and deteriorated lung function, it had extrapulmonary complications, such as cardiovascular problems, osteoporosis and muscle wasting. The concept of sarcopenia was proposed at first in 1989. It increases the risk of falls, disability and lowering life quality. Besides, it increased the mortality risk after admission from acute ward. Thereafter, sarcopenia is one of COPD co-morbidities, which should have great impacts of COPD. The studies showed sarcopenia reduced exercise capacities and worsening dyspnea scores. On the other hand, COPD exacerbation brings significant health burden. But there is limited data about the effect on sarcopenia on COPD exacerbation. We conducted a prospective observational study. We measured skeletal muscle mass and the strength of the used hand grip within 3 days of admission and before discharge. Mortality and exacerbation in one year are the primary end-points

ELIGIBILITY:
Inclusion criteria: Patients more than 45 years-old, were admitted due to COPD exacerbation.

COPD exacerbation criteria:

1. acute worsening respiratory symptoms without any other causes, And
2. Smoking more than 15 pack-years or the history of noxious gas exposure, And
3. Spirometry reports suggests obstructive ventilatory defect (FEV1/FVC <0.7) or
4. Attending physicians diagnose as COPD by clinical parameters if spirometry data are not available while enrolling.

Definite COPD exacerbation: fulfill 1、2、3 Probable COPD exacerbation: fulfill 1、2、4

Exclusion criteria:

1. Significant fluid retention such as edema, pleural effusion or ascites,
2. Patients with permanent pacemaker or implantable cardioverter defibrillator ,
3. Morbid obesity with BMI >34

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients more than 45 years-old, were admitted due to COPD exacerbation.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2020-06-21 (Actual)

PRIMARY OUTCOMES:
Mortality and exacerbations within 1 year of admission | 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author, [P.H.W], upon reasonable request

REFERENCES:
- [Derived] Lee CT, Wang PH. Handgrip strength during admission for COPD exacerbation: impact on further exacerbation risk. BMC Pulm Med. 2021 Jul 21;21(1):245. doi: 10.1186/s12890-021-01610-7. PMID 34289815